CLINICAL TRIAL: NCT06753929
Title: Assessment of Flow in Cerebrospinal Fluid Shunts with a Wireless Thermal Anisotropy Measurement Device During Routine Outpatient Surveillance Visits
Brief Title: Assessment of CSF Shunt Flow in an Outpatient Setting with a Thermal Measurement Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhaeos, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-06
Record Dates: First submitted 2024-12-09; First posted 2024-12-31 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Hydrocephalus
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- CSF Shunted Patients (Experimental): The trial will include two cohorts. The study device will be used to assess CSF flow in Cohort A (prospective). The study device will not be used for Cohort B (retrospective).
  Interventions: Device: wireless wearable thermal anisotropy measurement device

INTERVENTIONS:
Device: wireless wearable thermal anisotropy measurement device — non-invasive device used for assessing CSF shunt flow via thermal anisotropy measurements in a routine outpatient clinic setting

SUMMARY:
This study collects exploratory data using a non-invasive device for assessing CSF shunt flow using thermal anisotropy measurements. Patients with an existing implanted ventricular CSF shunt will be enrolled into either a prospective (study device) or retrospective (no study device) cohort to gather data on health resource utilization, quality-of-life, and study device measurements.

ELIGIBILITY:
Inclusion criteria

1. Existing ventricular cerebrospinal fluid shunt
2. Signed informed consent by subject or a parent, legal guardian, health care agent, or surrogate decision maker (according to local statutes)
3. Subject available for 2 week follow-up
4. Region of intact skin overlying an unambiguously identifiable palpable chronically indwelling ventricular shunt that crosses the clavicle; region of skin is appropriate in size for application of the study device (Cohort A only)

Exclusion Criteria

1. Presence of more than one distal shunt catheter in the study device measurement region
2. Presence of an interfering open wound or edema in the study device measurement region
3. Subject-reported history of serious adverse skin reactions to silicone-based adhesives
4. Participation in the study will interfere with, or be detrimental to, the administration of optimal health care to the subject

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 14 days
  Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health. A PROMIS T-score of 50 represents the general population norm, and each 10-point deviation represents one standard deviation from the norm. Higher scores equals more of the concept being measured (e.g., more Fatigue, more Physical Function).

CONTACTS AND LOCATIONS:
Locations (1):
- New Neurons Neurosurgical Institute, Cedar Knolls, New Jersey, United States